CLINICAL TRIAL: NCT04572867
Title: Efficacy of Aquapheresis in Patients Treated as Outpatients With Decompensated Heart Failure at a Veterans Hospital
Brief Title: Aquapheresis Efficacy in Outpatients With Decompensated Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low enrollment, COVID-19 pandemic causing suspension of most outpatient elective procedures, and no protected research time, Dr. Gelzer Bell is unable to continue this study.
Sponsor: Ramona Gelzer Bell (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Ramona Gelzer Bell, Director Congestive Heart Failure Program, James A. Haley Veterans Administration Hospital
Organization: James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AQUA
Record Dates: First submitted 2020-08-24; First posted 2020-10-01 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Heart Failure; Congestive Heart Failure; Decompensated Heart Failure
Keywords: Aquapheresis; Diuresis
MeSH Terms: conditions — Heart Failure | interventions — Ultrafiltration; Renal Dialysis; Diuretics

STUDY DESIGN:
Intervention Model Description: This is a Controlled Trial with two arms (aquapheresis and IV diuretics/Control), but there is the potential for cross-over to aquapheresis if a patient receiving diuretics is refractory to maximum doses of IV diuretics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Aquapheresis (Experimental): Per protocol, if randomized to Aquapheresis arm (AQ), all diuretics are discontinued and AQ will be administered as per established protocol. BMP and CBC will be checked prior to initiation and as needed, 7-10 days, 30, 60 and 90 days post discharge. Note, aquapheresis rate is to be decreased by 100 cc/hr if Hgb increases by 1gm/dL, and stopped if rate is decreased to 50 cc/hr or reaches euvolemia, whichever comes first.
  Interventions: Device: Aquapheresis
- IV Diuretics (Active Comparator): Per protocol (Fig 2), if randomized to IV diuretic therapy arm (IV), the patient will receive initial dose of IV diuretic based on base line renal function; then the dose will be doubled every 2 hrs if refractory, to a maximum of 8mg IV Bumex (or 320mg IV Lasix). Metolazone may be added at 2.5mg PO 30 minutes before loop diuretic if CR< 2.0, or 5mg PO if Cr > 2.0, if refractory to high dose loop diuretic. If a patient in IV arm is refractory to maximum 320 mg IV Lasix or 8 mg IV Bumex plus Metolazone then the patient may cross over to AQ arm.
  Interventions: Drug: IV Diuretics

INTERVENTIONS:
Device: Aquapheresis — The Aquadex FlexFlow® Fluid Removal System (from CHF Solutions™, Minneapolis, MN) is an FDA approved device that provides mechanical isosmotic fluid removal in volume-overloaded CHF patients via veno-venous ultrafiltration, and has been used in patients with congestive heart failure refractory to diuretics, it should be considered standard of care also. This study is using it in a randomized, controlled study in the Outpatient setting. The Aquadex FlexFlow® Fluid Removal System is a dual rotary pump device used with a sterile, single-use UF 500 Blood Circuit Set. Blood withdrawal is usually from a peripheral arm vein (such as the antecubital vein), using a 16 or 18- gauge, 3.5 cm catheter (similar to a standard IV catheter). A similar IV catheter is used for blood return via a second peripheral vein (typically in the forearm).
  Other Names: Ultrafiltration; Hemodialysis
  Arms: Aquapheresis
Drug: IV Diuretics — Active Comparator: Intravenous Diuretics Per protocol (Fig 2), if randomized to IV diuretic therapy arm (IV), the patient will receive initial dose of IV diuretic based on base line renal function; then the dose will be doubled every 2 hrs if refractory, to a maximum of 8mg IV Bumex (or 320mg IV Lasix). Metolazone may be added at 2.5mg PO 30 minutes before loop diuretic if CR< 2.0, or 5mg PO if Cr > 2.0, if refractory to high dose loop diuretic. If the patient in IV arm is refractory to max 320 mg IV Lasix or 8 mg IV Bumex plus Metolazone then the patient may cross over to AQ arm.
  Other Names: Intravenous Diuretics
  Arms: IV Diuretics

SUMMARY:
With this research the Investigators hope to learn if early aquapheresis in an outpatient setting will improve congestive heart failure symptoms in outpatients with decompensated heart failure who have been refractory to high dose diuretics. In previous trials in inpatient settings, aquapheresis has been demonstrated to improve quality of life and reduce hospital visits for those who have undergone the treatment. This study is one of the first to evaluate the effectiveness of aquapheresis in veterans with congestive heart failure in an outpatient setting.

The aquapheresis device, Aquadex FlexFlow® System, manufactured by CHF Solutions™, Minneapolis, MN, has been approved by the Food and Drug Administration (FDA) for removing excess sodium and fluid from patients suffering from volume overload, like in congestive heart failure.

DETAILED DESCRIPTION:
Congestive heart failure (CHF) affects nearly 2% of the U.S. population, with almost 1 million hospital admissions for acute decompensated CHF annually. Congestive heart failure is the most frequent cause of hospitalization in patients over the age of 65. Patients admitted for acute decompensated heart failure (ADHF) have a high 6-month readmission rate for acute CHF, ranging from 23% to 40% in different studies. It is estimated that 25 to 30% of these patients are diuretic resistant with 50% of patients losing less than 5 lbs. from admission weight and 20% actually gaining weight during the hospitalization.

Although loop diuretics have not been shown to improve survival in patients with CHF, they effectively alleviate symptoms of congestion. Diuretics have been part of standard CHF therapy in all recent survival trials of β-blockers, angiotensin converting enzyme inhibitors, and angiotensin II receptor blockers. Loop diuretics have been shown to be the most effective diuretics as single agents in moderate to severe heart failure. However, loop diuretics may be associated with increased morbidity and mortality attributable to deleterious effects on neurohormonal activation, electrolyte balance, and cardiac and renal function.

Removal of excessive fluid in patients with CHF is usually achieved by a combination of fluid and salt restriction and loop diuretics, but in some cases volume overload persists. Diuretic resistance is common, especially after chronic exposure to loop diuretics; patients require escalating doses (PO or IV to bypass delayed absorption in gut due to bowel edema), addition of another diuretic that works on different part of renal tubules (i.e. Thiazides) +/- diuretic drip and, if still refractory, ultimately Aquapheresis (a form of ultrafiltration).

Aquapheresis (AQ) compared to IV diuretics in the UNLOAD Trial (10), AQ safely produced greater weight loss, fluid removal, and reduction in 90-day readmission rate compared to IV diuretic. A meta-analysis of 10 randomized control trials (RCTs) showed AQ not only to be effective but safe. These observations suggest that a strategy of early ultrafiltration may improve responsiveness to diuretics, quicker weight loss, decrease hospitalization, readmission to hospital, ER or doctor visits with minimal risks. As result of these trials, American Hospital Association (AHA)/American College of Cardiology (ACC)/Heart Failure Society of American (HFSA) guidelines state it is reasonable to start Aquapheresis in patients with obvious volume overload or patients who are refractory to high dose diuretics (IIa, LOE B). Moreover, while this therapy is part of standard of care in an inpatient setting, many hospitals as a result of Affordable Care Act (ACA), have taken to AQ on an outpatient setting to further decrease the burden and attended cost associated with management of CHF. But the Investigators are unaware of any other prospective outpatient studies that have looked at the outcomes and cost effectiveness of aquapheresis.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be 18 years of age or older already on standard of care therapy including Angiotensin Converting Enzyme Inhibitors (ACE-I), Angiotensin

Receptor Blockers (ARBs), Sacubitril/Valsartan, beta-blocker, oral diuretic (80 mg Lasix/2 mg Bumex/40 mg Torsemide+/-Thiazide diuretic), and meet the following inclusion criteria to be enrolled:

Inclusion Criteria:

1. CHF refractory to oral diuretic (80mg Lasix, 2mg Bumex, or 40mg Torsemide)
2. Volume overload secondary to systolic or diastolic HF, evidenced by at least 2 of the following:

   1. Elevated BNP (>100)
   2. Paroxysmal nocturnal dyspnea or orthopnea
   3. Elevated jugular venous distention (>/ 7 cm)
   4. X-ray findings consisted with CHF
   5. Presence of ascites or LE edema . -

Exclusion Criteria:

1. Acute Coronary Syndrome
2. Hypertensive urgency or emergency
3. Rapid atrial fibrillation difficult to control
4. Contraindication to anticoagulation
5. Pregnancy
6. Requires hemodialysis (> CR > 3.0 mg/dl)
7. Symptomatic hypotension
8. Poor venous access
9. Pressor dependent. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Number of Hospitalizations by 7 days post-treatment | Between outpatient treatment and 7-days after outpatient treatment
  Compare number of hospitalization readmissions for CHF between Intervention (Aquaphersis arm) & Control groups
Number of Hospitalizations by 30 days post-treatment | Between outpatient treatment and 30 days after outpatient treatment
  Compare number of hospitalization readmissions for CHF between Intervention (Aquaphersis arm) & Control groups
Number of Hospitalizations by 60 days post-treatment | Between outpatient treatment and 60 days after outpatient treatment
  Compare number of hospitalization readmissions for CHF between Intervention (Aquaphersis arm) & Control groups
Number of Hospitalizations by 90 days post-treatment | Between outpatient treatment and 90 days after outpatient treatment
  Compare number of hospitalization readmissions for CHF between Intervention (Aquaphersis arm) & Control groups
Weight change by 7 days post-treatment | Outpatient treatment to 7 days after outpatient treatment
  Compare weight change (pounds) in patients between Intervention & Control groups
Weight change by 30 days post-treatment | Outpatient treatment to 30 days after outpatient treatment
  Compare weight change (pounds) in patients between Intervention & Control groups
Weight change by 60 days post-treatment | Outpatient treatment to 60 days after outpatient treatment
  Compare weight change (pounds) in patients between Intervention & Control groups
Weight change by 90 days post-treatment | Outpatient treatment to 90 days after outpatient treatment
  Compare weight change (pounds) in patients between Intervention & Control groups

SECONDARY OUTCOMES:
Total fluid removal | Baseline (Randomization) to outpatient discharge
  Compare total fluid removal (ml) in patients between Intervention & Control groups
Blood urea nitrogen at Baseline | Baseline (Randomization)
  Compare Blood urea nitrogen (BUN; mg/dl) (higher than normal range is worse) in patients between Intervention & Control groups
Blood urea nitrogen at 7 days post-treatment | 7 days after outpatient treatment
  Compare Blood urea nitrogen (BUN; mg/dl) (higher than normal range is worse) in patients between Intervention & Control groups
Blood urea nitrogen at 30 days post-treatment | 30 days after outpatient treatment
  Compare Blood urea nitrogen (BUN; mg/dl) (higher than normal range is worse)) in patients between Intervention & Control groups
Blood urea nitrogen at 60 days post-treatment | 60 days after outpatient treatment
  Compare Blood urea nitrogen (BUN; mg/dl) (higher than normal range is worse) in patients between Intervention & Control groups
Blood urea nitrogen at 90 days post-treatment | 90 days after outpatient treatment
  Compare Blood urea nitrogen (BUN; mg/dl) (higher than normal range is worse) in patients between Intervention & Control groups
Creatinine at Baseline | Baseline (Randomization)
  Compare Creatinine (Cr; mg/dl) (higher than normal range is worse) in patients between Intervention & Control groups
Creatinine at 7 days post-treatment | 7 days after outpatient treatment
  Compare Creatinine (Cr; mg/dl) (higher than normal range is worse) in patients between Intervention & Control groups
Creatinine at 30 days post-treatment | 30 days after outpatient treatment
  Compare Creatinine (Cr; mg/dl) (higher than normal range is worse) in patients between Intervention & Control groups
Creatinine at 60 days post-treatment | 60 days after outpatient treatment
  Compare Creatinine (Cr; mg/dl) (higher than normal range is worse) in patients between Intervention & Control groups
Creatinine at 90 days post-treatment | 90 days after outpatient treatment
  Compare Creatinine (Cr; mg/dl) (higher than normal range is worse) in patients between Intervention & Control groups
Glomerular filtration rate at Baseline | Baseline (Randomization)
  Compare Glomerular filtration rate (GFR; ml/min/1.73 meters squared) (lower than normal range is worse) in patients between Intervention & Control groups
Glomerular filtration rate at 7 days post-treatment | 7 days after outpatient treatment
  Compare Glomerular filtration rate (GFR; ml/min/1.73 meters squared) (lower than normal range is worse) in patients between Intervention & Control groups
Glomerular filtration rate at 30 days post-treatment | 30 days after outpatient treatment
  Compare Glomerular filtration rate (GFR; ml/min/1.73 meters squared) (lower than normal range is worse) in patients between Intervention & Control groups
Glomerular filtration rate at 60 days post-treatment | 60 days after outpatient treatment
  Compare Glomerular filtration rate (GFR; ml/min/1.73 meters squared) (lower than normal range is worse) in patients between Intervention & Control groups
Glomerular filtration rate at 90 days post-treatment | 90 days after outpatient treatment
  Compare Glomerular filtration rate (GFR; ml/min/1.73 meters squared) (lower than normal range is worse) in patients between Intervention & Control groups
Brain natriuretic peptide (BNP) test at Baseline | Baseline (Randomization)
  Compare BNP (pg/ml of blood) (higher than normal range is worse) in patients between Intervention & Control groups
Brain natriuretic peptide (BNP) test at 7 days post-treatment | 7 days after outpatient treatment
  Compare BNP (pg/ml of blood) (higher than normal range is worse) in patients between Intervention & Control groups
Brain natriuretic peptide (BNP) test at 30 days post-treatment | 30 days after outpatient treatment
  Compare BNP (pg/ml of blood) (higher than normal range is worse) in patients between Intervention & Control groups
Brain natriuretic peptide (BNP) test at 60 days post-treatment | 60 days after outpatient treatment
  Compare BNP (pg/ml of blood) (higher than normal range is worse) in patients between Intervention & Control groups
Brain natriuretic peptide (BNP) test at 90 days post-treatment | 90 days after outpatient treatment
  Compare BNP (pg/ml of blood) (higher than normal range is worse) in patients between Intervention & Control groups
6-minute Walk Test at Baseline | Baseline (Randomization)
  Compare 6-minute Walk Test (meters/6 minutes; less distance means more disability) in patients between Intervention & Control groups
6-minute Walk Test at 7 days post-treatment | 7 days after outpatient treatment
  Compare 6-minute Walk Test (meters/6 minutes; less distance means more disability) in patients between Intervention & Control groups
6-minute Walk Test at 30 days post-treatment | 30 days after outpatient treatment
  Compare 6-minute Walk Test (meters/6 minutes; less distance means more disability) in patients between Intervention & Control groups
6-minute Walk Test at 60 days post-treatment | 60 days after outpatient treatment
  Compare 6-minute Walk Test (meters/6 minutes; less distance means more disability) in patients between Intervention & Control groups
6-minute Walk Test at 90 days post-treatment | 90 days after outpatient treatment
  Compare 6-minute Walk Test (meters/6 minutes; less distance means more disability) in patients between Intervention & Control groups
Minnesota Living with Heart Failure Questionnaire (MLWHFQ) | Baseline (Randomization)
  Compare Minnesota Living with Heart Failure Questionnaire (MLWHFQ) (total score; higher score means more impairment) in patients between Intervention & Control groups
Minnesota Living with Heart Failure Questionnaire (MLWHFQ) | 7 days after outpatient treatment
  Compare Minnesota Living with Heart Failure Questionnaire (MLWHFQ) (total score; higher score means more impairment) in patients between Intervention & Control groups
Minnesota Living with Heart Failure Questionnaire (MLWHFQ) | 30 days after outpatient treatment
  Compare Minnesota Living with Heart Failure Questionnaire (MLWHFQ) (total score; higher score means more impairment) in patients between Intervention & Control groups
Minnesota Living with Heart Failure Questionnaire (MLWHFQ) | 60 days after outpatient treatment
  Compare Minnesota Living with Heart Failure Questionnaire (MLWHFQ) (total score; higher score means more impairment) in patients between Intervention & Control groups
Minnesota Living with Heart Failure Questionnaire (MLWHFQ) | 90 days after outpatient treatment
  Compare Minnesota Living with Heart Failure Questionnaire (MLWHFQ) (total score; higher score means more impairment) in patients between Intervention & Control groups
SF-36 at Baseline | Baseline (Randomization)
  Compare SF-36 weighted sums (0-100 scale; lower score means more disability) in patients between Intervention & Control groups
SF-36 at 7 days post-treatment | 7 days after outpatient treatment
  Compare SF-36 weighted sums (0-100 scale; lower score means more disability) in patients between Intervention & Control groups
SF-36 at 30 days post-treatment | 30 days after outpatient treatment
  Compare SF-36 weighted sums (0-100 scale; lower score means more disability) in patients between Intervention & Control groups
SF-36 at 60 days post-treatment | 60 days after outpatient treatment
  Compare SF-36 weighted sums (0-100 scale; lower score means more disability) in patients between Intervention & Control groups
SF-36 at 90 days post-treatment | 90 days after outpatient treatment
  Compare SF-36 weighted sums (0-100 scale; lower score means more disability) in patients between Intervention & Control groups
Adverse events: bleeding incidents during Outpatient treatment | Start of treatment to discharge, which is usually the same day, but up to 3 days post-treatment, if medically necessary.
  Compare number of Adverse Events (bleeding incidents) in patients between Intervention & Control groups: bleeding, line-related infection, etc.
Adverse events: line infections during Outpatient treatment | Start of treatment to up to 14 days post-treatment.
  Compare number of Adverse Events (line infections) in patients between Intervention & Control groups: bleeding, line-related infection, etc.
Costs | Baseline (Randomization) to 90 days post-discharge
  Compare costs (dollars) between Intervention & Control groups

CONTACTS AND LOCATIONS:
Overall Officials: Ramona Gelzer Bell, MD, Principal Investigator — James A. Haley Veterans Administration Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polanczyk CA, Newton C, Dec GW, Di Salvo TG. Quality of care and hospital readmission in congestive heart failure: an explicit review process. J Card Fail. 2001 Dec;7(4):289-98. doi: 10.1054/jcaf.2001.28931. PMID 11782850
- [Background] Hamner JB, Ellison KJ. Predictors of hospital readmission after discharge in patients with congestive heart failure. Heart Lung. 2005 Jul-Aug;34(4):231-9. doi: 10.1016/j.hrtlng.2005.01.001. PMID 16027642
- [Background] Krumholz HM, Chen YT, Wang Y, Vaccarino V, Radford MJ, Horwitz RI. Predictors of readmission among elderly survivors of admission with heart failure. Am Heart J. 2000 Jan;139(1 Pt 1):72-7. doi: 10.1016/s0002-8703(00)90311-9. PMID 10618565
- [Background] Lee WY, Capra AM, Jensvold NG, Gurwitz JH, Go AS; Epidemiology, Practice, Outcomes, and Cost of Heart Failure (EPOCH) Study. Gender and risk of adverse outcomes in heart failure. Am J Cardiol. 2004 Nov 1;94(9):1147-52. doi: 10.1016/j.amjcard.2004.07.081. PMID 15518609
- [Background] Adams KF Jr, Fonarow GC, Emerman CL, LeJemtel TH, Costanzo MR, Abraham WT, Berkowitz RL, Galvao M, Horton DP; ADHERE Scientific Advisory Committee and Investigators. Characteristics and outcomes of patients hospitalized for heart failure in the United States: rationale, design, and preliminary observations from the first 100,000 cases in the Acute Decompensated Heart Failure National Registry (ADHERE). Am Heart J. 2005 Feb;149(2):209-16. doi: 10.1016/j.ahj.2004.08.005. PMID 15846257
- [Background] Consensus recommendations for the management of chronic heart failure. On behalf of the membership of the advisory council to improve outcomes nationwide in heart failure. Am J Cardiol. 1999 Jan 21;83(2A):1A-38A. No abstract available. PMID 10072251
- [Background] Wilcox CS. Diuretics. In: Brenner BM, Rector FC. The kidney. Philadelphia: WB Saunders, 1996: 2299-330.
- [Background] Ellison DH. Diuretic therapy and resistance in congestive heart failure. Cardiology. 2001;96(3-4):132-43. doi: 10.1159/000047397. PMID 11805380
- [Background] Schrier RW. Role of diminished renal function in cardiovascular mortality: marker or pathogenetic factor? J Am Coll Cardiol. 2006 Jan 3;47(1):1-8. doi: 10.1016/j.jacc.2005.07.067. Epub 2005 Dec 15. PMID 16386657
- [Background] Costanzo MR, Guglin ME, Saltzberg MT, Jessup ML, Bart BA, Teerlink JR, Jaski BE, Fang JC, Feller ED, Haas GJ, Anderson AS, Schollmeyer MP, Sobotka PA; UNLOAD Trial Investigators. Ultrafiltration versus intravenous diuretics for patients hospitalized for acute decompensated heart failure. J Am Coll Cardiol. 2007 Feb 13;49(6):675-83. doi: 10.1016/j.jacc.2006.07.073. Epub 2007 Jan 26. PMID 17291932
- [Background] Sharma A, Hermann DD, Mehta RL. Clinical benefit and approach of ultrafiltration in acute heart failure. Cardiology. 2001;96(3-4):144-54. doi: 10.1159/000047398. PMID 11805381
- [Background] Marenzi G, Lauri G, Grazi M, Assanelli E, Campodonico J, Agostoni P. Circulatory response to fluid overload removal by extracorporeal ultrafiltration in refractory congestive heart failure. J Am Coll Cardiol. 2001 Oct;38(4):963-8. doi: 10.1016/s0735-1097(01)01479-6. PMID 11583865
- [Background] Rimondini A, Cipolla CM, Della Bella P, Grazi S, Sisillo E, Susini G, Guazzi MD. Hemofiltration as short-term treatment for refractory congestive heart failure. Am J Med. 1987 Jul;83(1):43-8. doi: 10.1016/0002-9343(87)90495-5. PMID 3605181
- [Background] Jaski BE, Ha J, Denys BG, Lamba S, Trupp RJ, Abraham WT. Peripherally inserted veno-venous ultrafiltration for rapid treatment of volume overloaded patients. J Card Fail. 2003 Jun;9(3):227-31. doi: 10.1054/jcaf.2003.28. PMID 12815573
- [Background] Agostoni P, Marenzi G, Lauri G, Perego G, Schianni M, Sganzerla P, Guazzi MD. Sustained improvement in functional capacity after removal of body fluid with isolated ultrafiltration in chronic cardiac insufficiency: failure of furosemide to provide the same result. Am J Med. 1994 Mar;96(3):191-9. doi: 10.1016/0002-9343(94)90142-2. PMID 8154506
- [Background] Liang KV, Hiniker AR, Williams AW, Karon BL, Greene EL, Redfield MM. Use of a novel ultrafiltration device as a treatment strategy for diuretic resistant, refractory heart failure: initial clinical experience in a single center. J Card Fail. 2006 Dec;12(9):707-14. doi: 10.1016/j.cardfail.2006.08.210. PMID 17174232
- [Background] Kwok CS, Wong CW, Rushton CA, Ahmed F, Cunnington C, Davies SJ, Patwala A, Mamas MA, Satchithananda D. Ultrafiltration for acute decompensated cardiac failure: A systematic review and meta-analysis. Int J Cardiol. 2017 Feb 1;228:122-128. doi: 10.1016/j.ijcard.2016.11.136. Epub 2016 Nov 9. PMID 27863352
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Heart Failure Society of America; Lindenfeld J, Albert NM, Boehmer JP, Collins SP, Ezekowitz JA, Givertz MM, Katz SD, Klapholz M, Moser DK, Rogers JG, Starling RC, Stevenson WG, Tang WH, Teerlink JR, Walsh MN. HFSA 2010 Comprehensive Heart Failure Practice Guideline. J Card Fail. 2010 Jun;16(6):e1-194. doi: 10.1016/j.cardfail.2010.04.004. PMID 20610207
- [Background] Kazory A. Ultrafiltration Therapy for Heart Failure: Balancing Likely Benefits against Possible Risks. Clin J Am Soc Nephrol. 2016 Aug 8;11(8):1463-1471. doi: 10.2215/CJN.13461215. Epub 2016 Mar 31. PMID 27034400
- [Background] Jain A, Agrawal N, Kazory A. Defining the role of ultrafiltration therapy in acute heart failure: a systematic review and meta-analysis. Heart Fail Rev. 2016 Sep;21(5):611-9. doi: 10.1007/s10741-016-9559-2. PMID 27154520
- [Background] Costanzo MR, Ronco C, Abraham WT, Agostoni P, Barasch J, Fonarow GC, Gottlieb SS, Jaski BE, Kazory A, Levin AP, Levin HR, Marenzi G, Mullens W, Negoianu D, Redfield MM, Tang WHW, Testani JM, Voors AA. Extracorporeal Ultrafiltration for Fluid Overload in Heart Failure: Current Status and Prospects for Further Research. J Am Coll Cardiol. 2017 May 16;69(19):2428-2445. doi: 10.1016/j.jacc.2017.03.528. PMID 28494980
- [Background] Kazory A, Costanzo MR. Extracorporeal Isolated Ultrafiltration for Management of Congestion in Heart Failure and Cardiorenal Syndrome. Adv Chronic Kidney Dis. 2018 Sep;25(5):434-442. doi: 10.1053/j.ackd.2018.08.007. PMID 30309461